CLINICAL TRIAL: NCT05225675
Title: A Phase 2, Randomized, Double-Blinded, Placebo-Controlled, Parallel-Group, Multicenter Trial to Evaluate the Safety and Tolerability, Efficacy, Pharmacokinetics, Pharmacodynamics, and Immunogenicity of 2 Dose Regimens of ARGX-117 in Adults with Multifocal Motor Neuropathy
Brief Title: A Clinical Trial to Investigate the Safety and Tolerability, Efficacy, Pharmacokinetics, Pharmacodynamics and Immunogenicity of 2 Dose Regimens of ARGX-117 in Adults with Multifocal Motor Neuropathy
Acronym: ARDA
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: argenx (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ARGX-117-2002
Record Dates: First submitted 2021-11-05; First posted 2022-02-04 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Multifocal Motor Neuropathy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- ARGX-117 (Experimental): Intravenous administration of ARGX-117
  Interventions: Biological: ARGX-117
- Placebo (Placebo Comparator): Intravenous administration of placebo
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: ARGX-117 — Intravenous administration of ARGX-117
  Arms: ARGX-117
Other: Placebo — Intravenous administration of placebo
  Arms: Placebo

SUMMARY:
This is a phase 2, randomized, double-blinded, placebo-controlled, parallel-group, multicenter trial to evaluate the safety and efficacy of 2 dose regimens of ARGX-117 versus placebo, in participants with MMN previously stabilized with IVIg (intravenous immunoglobulin).

ELIGIBILITY:
Inclusion Criteria:

1. Capable of giving signed informed consent form (ICF)
2. Male/female at least 18 years of age at the time the informed consent form (ICF) is signed
3. Probable or definite MMN according to the European Federation of Neurological Societies (EFNS)/Peripheral Nerve Society (PNS) (EFNS/PNS) 2010 guidelines at screening confirmed by the MMN Confirmation Committee (MCC)
4. Receiving a stable IVIg regimen for at least 3 months before screening or recently initiated IVIg treatment
5. IVIg treatment dependency confirmation by the MMN Confirmation Committee (MCC)
6. Immunization with the first meningococcal vaccine and pneumococcal vaccine, and the single Haemophilus influenza type B vaccine must be performed at least 14 days before IMP administration at V1 according to local country-specific immunization schedules. A documented history of vaccination against Neisseria meningitides, Haemophilus influenza type B, and streptococcus pneumonia will be permitted
7. Contraceptive use by men and women should be consistent with local regulations regarding the methods of contraception for those participating in clinical studies

Exclusion Criteria:

1. Any coexisting condition which may interfere with the outcome assessments
2. Clinical signs or symptoms suggestive for neuropathies other than MMN such as motor neuron disease or other inflammatory neuropathies
3. Severe psychiatric disorder, history of suicide attempt, or current suicidal ideation that in the opinion of the investigator could create undue risk to the participant or could affect adherence with the trial protocol.
4. Clinically significant uncontrolled active or chronic bacterial, viral, or fungal infection during the screening and/or IVIg monitoring period (IVMP).
5. Any other known autoimmune disease that, in the opinion of the investigator, would interfere with an accurate assessment of clinical symptoms of MMN or put the participant at undue risk (eg, SLE).
6. History of malignancy unless resolved by adequate treatment with no evidence of recurrence for ≥3 years before the first administration of the IMP. Participants with the following carcinomas will be eligible:

   1. Adequately treated basal cell or squamous cell skin cancer
   2. Carcinoma in situ of the cervix
   3. Carcinoma in situ of the breast
   4. Incidental histological finding of prostate cancer
7. Clinical evidence of other significant serious diseases, have had a recent major surgery (including a splenectomy at any time), or who have any other condition in the opinion of the investigator, that could confound the results of the trial or put the participant at undue risk
8. Prior/concomitant therapy

   1. Cyclophosphamide and/or rituximab and/or eculizumab and/or mycophenolate mofetil within 3 months prior to screening
   2. Use of an investigational product within 3 months or 5 half-lives (whichever is longer) before the first dose of the IMP.
9. Positive serum test at screening for an active viral infection with any of the following conditions:

   1. Hepatitis B virus (HBV) that is indicative of an acute or chronic infection
   2. Hepatitis C virus (HCV) based on HCV antibody assay
   3. HIV based on test results that are associated with an AIDS-defining condition
10. Current or history of (ie, within 12 months of screening) alcohol, drug, or medication abuse
11. Known hypersensitivity reaction to 1 of the components of the IMP or any of its excipients
12. Female participants with a positive serum or urine pregnancy test, lactating females, and those who intend to become pregnant during the trial or within 15 months after last dose of the IMP
13. ALT or AST ≥2 × upper limit of normal and total bilirubin ≥1.5 × upper limit of normal of the central laboratory reference range
14. An estimated glomerular filtration rate of ≤60 mL/min/1.73m2

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2022-03-31 (Actual); Primary Completion 2024-06-04 (Actual); Study Completion 2024-06-04 (Actual)

PRIMARY OUTCOMES:
Safety outcomes based on adverse event (AE) monitoring and other safety assessments | 16 weeks

SECONDARY OUTCOMES:
Time to the first retreatment with IVIg since the final IVIg treatment of the IVIg monitoring period | 16 weeks
AUC (area under curve) of the change from baseline in mMRC (modified Medical Research Council)-10 sum score | 16 weeks
Change from baseline in the average score of the 2 most important muscle groups as assessed by the mMRC (modified Medical Research Council)-14 sum score | 16 weeks
Value baseline in the mMRC (modified Medical Research Council)-14 sum score | 16 weeks
Change from baseline in the mMRC (modified Medical Research Council)-14 sum score | 16 weeks
Proportion of participants showing a deterioration of 1 or more points in at least 2 muscle groups as assessed by the mMRC (modified Medical Research Council)-14 sum score | 16 weeks
Proportion of participants with no deterioration in 2 or more muscle groups as assessed by mMRC (modified Medical Research Council)-14 sum score | 16 weeks
AUC (area under curve) of the change from baseline in GS (grip strength) | 16 weeks
Proportion of participants with a GS (grip strength) decrease of 8 kilopascal (kPa) or more over 3 consecutive days | 16 weeks
Values baseline in GS (grip strength) | 16 weeks
  The baseline for the grip strength is a 3-day moving average per hand, measured as an average of 3 contractions daily, each lasting 3 seconds.
  Measurement of GS will be done using the Martin vigorimeter in kPa.
Change from baseline in GS (grip strength) | 16 weeks
  The baseline for the grip strength is a 3-day moving average per hand, measured as an average of 3 contractions daily, each lasting 3 seconds.
  Measurement of GS will be done using the Martin vigorimeter in kPa.
Percent change from baseline in GS (grip strength) | 16 weeks
  The baseline for the grip strength is a 3-day moving average per hand, measured as an average of 3 contractions daily, each lasting 3 seconds.
  Measurement of GS will be done using the Martin vigorimeter in kPa.
Values baseline in the Rasch-built overall disability scale for MMN (MMN-RODS©) | 16 weeks
Change from baseline in the Rasch-built overall disability scale for MMN (MMN-RODS©) | 16 weeks
Values baseline in the average time for upper extremity (arm and hand) function (9-Hole Peg Test [9-HPT], or timed Peg Board Test) | 16 weeks
Change from baseline in the average time for upper extremity (arm and hand) function (9-Hole Peg Test [9-HPT], or timed Peg Board Test) | 16 weeks
Proportion of participants by level of severity on each dimension of the EQ-5D-5L scale | 16 weeks
Change from baseline in quality of life using EQ-5D-5L visual analog scale | 16 weeks
Change from baseline in the chronic acquired polyneuropathy patient-reported index (CAP-PRI) | 16 weeks
Serum titer levels of binding antibodies (BAbs) against ARGX-117 | 16 weeks
Change from baseline in free C2, total C2, functional complement activity (CH50) | 16 weeks
Values baseline in free C2, total C2, functional complement activity (CH50) | 16 weeks
Area Under The Curve (AUC) | 16 weeks
Maximum serum concentrations (Cmax) | 16 weeks

CONTACTS AND LOCATIONS:
Locations (40):
- United States (13):
  - HonorHealth Research Institute-Neuroscience Research, Scottsdate, Arizona
  - California Pacific Medical Center-Forbes Norris MDA/ALS Research Center, San Francisco, California
  - George Washington Medical Faculty Associates, Washington D.C., District of Columbia
  - HonorHealth Research Institute-Neuroscience Research, Maitland, Florida
  - University of South Florida Carol and Frank Morsani Center for Advanced Healthcare, Tampa, Florida
  - NorthShore University HealthSystem, Glenview, Illinois
  - University of Kansas Medical Center, Kansas City, Kansas
  - University of Minnesota Delware Clinic Research Unit, Minneapolis, Minnesota
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - Perelman Center for Advanced Medicine-University of Penssylvania, Philadelphia, Pennsylvania
  - Austin Neuromuscular Center, Austin, Texas
  - West Virginia University Medicine, Morgantown, West Virginia
- Medizinische Universitat Wien Universitatsklienik fur Neurologie, Vienna, Austria
- AZ Sint-Lucas, Ghent, Belgium
- Canada (2):
  - Genge Partners Montreal, Québec
  - Toronto General Hospital, Toronto
- France (4):
  - CHU de Bordeaux-Hopital Pellegrin, Bordeaux
  - CHRU de Lille-Hopital Roger Salengro, Lille
  - CHU de Nice-Hopital Pasteur 2, Nice
  - Hopital Pitie Salpetriere, Paris
- Germany (5):
  - Katholisches Klinikum Bochum, Bochum
  - Universitatsklinikum Essen, Essen
  - Universitatsmedzin Gottingen, Klinik fur Neurologie, Göttingen
  - Medizinische Hochschule Hannover Klinik Fur Neurologie, Hanover
  - Universitatsklinikum Munster, Münster
- Italy (4):
  - IRCCS Ospedale San Raffaele, Milan
  - Azienda Ospedaliero Univeritaria Pisana-UOS Neurologia, Pisa
  - Azienda Ospedaliera Sant'Andrea-UOS Malattie Neuromuscolari, Rome
  - Instituto Clinico Humanitas (IRCCS), Rozzano
- Netherlands (2):
  - Amsterdam UMC location AMC, Dep of Neurology, Amsterdam
  - University Medical Centre Utrecht, Utrecht
- Poland (2):
  - Michalscy I Partnerzy Lekarze Spolka Partnerska, Krakow
  - Uniwersyteckie centrum kliniczne Warszawskiego, Warsaw
- Spain (3):
  - Hospital Universitario Vall d'Herbon, Barcelona
  - Hospital de la Santa Creu I Santa Pau -Sevicio Neurologia, Barcelona
  - Hospital Universitari I Politecnic La Fe de Valencia-Servicio Neurologia, Valencia
- United Kingdom (3):
  - Queen Elisabeth University Hospital, Glasgow
  - University College London Hospital, London
  - Oxford University Hospitals NHS Trust-Jonh Radcliffe Hospital, Oxford

IPD SHARING:
Plan to Share IPD: No